CLINICAL TRIAL: NCT00172172
Title: A Study to Evaluate the Effects of Calcium Supplementation on the Efficacy and Safety of Recombinant Human Parathyroid Hormone (ALX1-11) in Postmenopausal Women With Osteoporosis (CAP Study)
Brief Title: Calcium Supplementation in Postmenopausal Women
Acronym: CAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL1-11-008
Expanded Access: Available
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Osteoporosis
Keywords: Post-menopausal; Osteoporosis; Parathyroid Hormone; PTH; ALX1-11
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): PTH 100 mcg and 700 mg calcium
  Interventions: Drug: PTH/Calcium
- 2 (Experimental): PTH 100 mcg and placebo
  Interventions: Drug: PTH/placebo
- 3 (Placebo Comparator): Placebo and 700 mg calcium
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: PTH/Calcium — PTH(1-84) subcutaneous injection and calcium 700 mg oral
  Other Names: PREOS
  Arms: 1
Drug: PTH/placebo — PTH (1-84) injected subcutaneously and placebo provided orally
  Other Names: PREOS
  Arms: 2
Drug: placebo — Placebo injected subcutaneously and 700 mg calcium orally
  Arms: 3

SUMMARY:
This study is evaluating the effects of calcium supplementation on the efficacy and safety of recombinant parathyroid hormone (ALX1-11) in postmenopausal women with osteoporosis. The primary objective of this clinical study is to evaluate whether increases in bone mineral density (BMD) for subjects treated with ALX1-11 and receiving no calcium supplementation are less than increases in BMD observed for subjects treated with ALX1-11 and receiving calcium supplementation.

DETAILED DESCRIPTION:
Effects of ALX1-11 on bone mineral density (BMD) have been documented in a dose-finding Phase II clinical trial in osteoporotic postmenopausal women, supplemented with calcium and Vitamin D3 but without any other treatment for osteoporosis. The anabolic effects of ALX1-11 in the lumbar vertebrae were statistically significant after the 12-month treatment period and more pronounced than any approved therapy. Additionally, animal studies have shown that the new bone formed by treatment with ALX1 11 is of good quality both histologically and biomechanically.

The primary objective of this clinical study is to evaluate whether increases in bone mineral density (BMD) for subjects treated with ALX1-11 and receiving no calcium supplementation are less than increases in BMD observed for subjects treated with ALX1-11 and receiving calcium supplementation.

A secondary objective of this clinical study are to evaluate whether changes in other efficacy parameters, such as bone mineral content (BMC) and biochemical markers of bone turnover, for subjects treated with ALX1-11 and receiving no calcium supplementation are less than increases observed for subjects treated with ALX1-11 and receiving calcium supplementation.

This is a double-blind, multi-centered, randomized, placebo-controlled, parallel-group study comprised of 3 treatment groups: ALX1-11 injection plus oral calcium, ALX1-11 injection plus oral placebo calcium, and placebo ALX1-11 injection plus oral calcium. All subjects also receive 400 IU oral vitamin D3. The dose of ALX1-11 to be used in this study is 100 μg, self administered by daily sc injection. The calcium dose is 700 mg/day.

Additional supplemental calcium and/or Vitamin D3 will not be permitted. Patients will be monitored for the development of hypercalcemia and/or hypercalciuria.

ELIGIBILITY:
Inclusion Criteria:

* Women who are capable of understanding and giving written, voluntary informed consent before the clinical study screening visit
* Women with the ability to self-administer a daily injection or having a designee who will give the injections
* Women who are postmenopausal with at least one year since their last menstruation. If a subject's menopausal status at screening is in question, because of history or because the subject had a hysterectomy without oophorectomy, a follicle-stimulating hormone (FSH) level >40 mIU/mL will satisfy the definition of postmenopausal status.
* Women 45-54 years of age with the following T-score and/or vertebral fracture

  * T-score >=3.0 standard deviations (SD) below mean peak bone mass of young women at the lumbar spine, femoral neck, or total hip Or
  * T-score >=2.5 SD below mean peak bone mass of young women at the lumbar spine, femoral neck, or total hip with a prevalent vertebral fracture verified by the central imaging organization before the subject is enrolled into the study
* Women >=55 years of age with the following T-score and/or vertebral fracture:

  o T-score >=2.5 SD below mean peak bone mass of young women at the lumbar spine, femoral neck, or total hip Or
* T-score >=2.0 SD below mean peak bone mass of young women at the lumbar spine, femoral neck, or total hip with a vertebral fracture verified by the central imaging organization before the subject is enrolled into the study

The following types of vertebral fractures should not be considered for subject enrollment into this study:

* Pathological fractures due to malignant disease or infection
* Fractures due to excessive trauma sufficient to cause a fracture in young individuals with normal bone mass

Exclusion Criteria:

A. Vertebral Deformity (assessed as described in Appendix 2 of the protocol, are sufficient for exclusion):

· Vertebral deformities

* Patient has 5 or more vertebral (thoracic and lumbar) fractures
* Patient has 2 or more lumbar vertebral deformities (L1 to L4)

B. DXA Imaging:

· Inability to have a DXA scan performed, e.g.:

* A history of a lumbar laminectomy which interferes with the DXA measurement of the lumbar vertebrae
* The presence of pedicle screws
* The patient cannot lay flat on her back for the required time to provide accurate imaging
* Patient is not able to have an A/P lumbar vertebral DXA performed
* Patient has a history of vertebroplasty
* Any other excessive degenerative disease which interferes with the DXA measurement of the lumbar vertebrae or hip

C. History of or Concurrent Illness:

* Disorders of Immunity

  * HIV
  * Significant* immunological disorders
* Endocrine system

  * Any history of hyper- or hypoparathyroidism
  * Cushing's disease
  * Hyperthyroidism (within 12 months)
  * Significant* endocrine disorders
* Gastrointestinal system

  - Significant* gastrointestinal disorders
* Kidney and collecting system

  * Clinically significant* history of nephrolithiasis or urolithiasis
  * Current impaired renal function and/or verified kidney calcification*
  * Significant* renal disorders
* Liver, biliary tract and pancreatic systems

  * Active hepatitis or pancreatitis
  * Significant* hepatic or pancreatic disorders
* Musculoskeletal system

  * Any history of other metabolic bone diseases within the past 5 years, (e.g., Paget´s disease, osteogenesis imperfecta, osteomalacia)
  * Subjects with chronic, active joint disease and/or joint infection
* Neoplasia - Any history of bone cancer or any cancer within the previous 5 years, with the exception of squamous or basal cell carcinoma**

(**)Patients who have had either squamous or basal cell carcinoma of the skin can enroll if:

1. The lesion(s) were fully resected with clear margins described in a written report by a pathologist, and
2. The patient has had no recurrence of lesions for at least one year from the time of the original resection.

   · Nervous system
   * Significant* neurological or psychiatric disease

     · Vascular, respiratory and cardiac system
   * Significant* unstable cardiac or pulmonary disease

   (*) Significance will be determined by the investigator on the basis of history, physical exam, and/or laboratory screens. Significant disorders necessitate ongoing changes in therapeutic medication or frequent monitoring.

   D. Concurrent Medication:

   Patients cannot be enrolled into this clinical trial if they have received any of the following therapies at any time:
   * Any PTH or PTH analogs [e.g., rhPTH(1-84), PTH(1-34), PTHrP and analogs]
   * Fluoride
   * Strontium

   Patients must have been off the following agents for the specified times before entering the screening phase of this clinical trial:
   * Any investigational drug (>30 days)
   * Anabolic steroids or androgens (>6 consecutive months)
   * Active Vitamin D3 metabolites and analogs, e.g., calcitriol (>90 days)
   * Provera (medroxyprogesterone) (According to label instructions)
   * Systemic corticosteroids, more than 5mg/day formulation equivalent to 5mg/day prednisone (>12 consecutive month or as acute bolus for nonrecurring condition). A patient who has been enrolled in the study and needs to receive an acute bolus of steroids (oral or injectable) for a self-limited illness may continue treatment in the study if the following requirements are met:

     * The maximal dose of steroid (prednisone equivalent) is limited to no more than 225 mg (7.5 mg each day for 30 days)
     * The illness is acute in nature and is not expected to recur during the remaining treatment period of the study
   * Inhaled corticosteroids equivalent to <1200 μg of beclomethasone
   * Bisphosphonates, including investigational bisphosphonates

     * If the patient has received bisphosphonates for >90 days during 12 months immediately before screening, the patient is excluded from this study.
     * If the patient has received bisphosphonates for more than 12 months at any time.

       *The patient may be enrolled if she:

   Has taken bisphosphonates for >=30 days but <=90 days, and has completed washout of equivalent time.

   No washout is necessary if the patient has taken bisphosphonates <30 days.
   * Intravenous (IV) pamidronate

     * Patient can have received 1 dose of pamidronate in >3 to 12 months immediately preceding the screening visit. Patient should not have received this 1 dose within the three months immediately prior to the screening visit
     * Patient must not have received >2 doses at any time before screening.
   * Cyclical Etidronate

     * Patient should not have an exposure equal to 9 months on a standard dose (e.g., 400 mg).
     * Exposure to cyclical etidronate must be <=6 months on a standard dose (e.g., 400 mg/day) prior to the screening visit.
   * Phenytoin for seizure control:

     * If the patient has received phenytoin <5 years before, the patient is excluded from this study

       * The patient may continue in the screening process if:

   >=15 years have passed since the last dose of phenytoin or if use was between 5-15 years before the screening visit and the patient received phenytoin for <2 months

   Patients may be enrolled if they have been stabilized on the following therapy for the specified amount of time:
   * Thyroid Hormone (<0.1 mg/day thyroxine) therapy for >=6 months

     - If taking >= 0.1 mg/day but <= 0.2 mg/day, must have serum TSH level >= 0.1 mU/L. Patients will be excluded if they are taking doses of >0.2 mg/day.
     * If a patient has had a minimal change in L-thyroxine dose of <=0.025 mg/day within 6 months of enrollment, and has been on this new dose for >=2 months, she may continue. The patient must have the history documented with L-thyroxine in the CRF.
     * If a patient requires an increase or decrease in her thyroid replacement dose, after she has been enrolled in this clinical study, each increment or decrement should be <=0.025 mg/day, and increments should not occur more frequently than once per month, as recommended by a physician who is caring for the patient. The patient must have a TSH and thyroxine level within 3 months of the dose change to ensure that the patient does not become hyperthyroid, or hypothyroid.
   * Thiazide (Stable dosage of thiazide for >=3 consecutive months)

   All patients must stop the following therapies at least 4 weeks before starting the stabilization period and will remain off these therapies for the remainder of the clinical study. The informed consent must be signed prior to the washout of any therapy. Screening laboratories must be performed only after the washout is complete. However, imaging studies (BMD, X-rays) may be performed prior to starting the calcitonin, estrogen, or Selective Estrogen Receptor Modulation (SERM) washout.

   · Calcitonin
   * Estrogen replacement therapy by oral, transdermal, or intramuscular administration
   * Vaginal application of estrogen-containing creams (If conjugated estrogen or estradiol: <=0.5 g twice each week [total of 1.0 g weekly] this medication is allowed)
   * SERM drugs, e.g., tamoxifen, raloxifene, Evista
   * Cytostatics, e.g., azathioprine, recombinant human tumor necrosis fusion (Fc) protein, monoclonal antibody against tumor necrosis factor (e.g., remicade [infliximab]
   * Medication known to affect the metabolism of bone (the Principal Investigator should discuss this with the PMO before the patient is excluded from enrollment).

   E. Miscellaneous Concurrent Medications

   · Methotrexate,which interferes with DNA synthesis, repair and cellular replication.

   · Immunomodulatory agents with antiproliferative activity.

   · Intra-articular injections

   - Patients may receive a maximum of 1 intra-articular injection (ONE JOINT ONLY) every 6 months while participating in this study. The dose of corticosteroid injected should not exceed the anti-inflammatory equivalent dose of Prednisone 40-mg suspension. The dose and volume should be adjusted downward as appropriate to the size of the joint.

   F. Laboratory Values and Physical Examination Findings:

   -For laboratory values, the levels shown below are the upper limits for exclusions based on specific test results. For weight, the limit is the lower limit.

   · Serum calcium >10.7 mg/dL (>2.67 mmol/L)

   · Serum creatinine > 1.5 mg/dL (132.6 µmol/L)

   · Urinary calcium to creatinine ratio >=1.0 (mmol/mmol)
   * Total serum alkaline phosphatase >130 U/L (Serum total alkaline phosphatase value given is for the U.S.; >311 U/L (Argentina), >159 U/L (Mexico).
   * Body weight <40 kg

   G. Substance Abuse:

   · Subjects are excluded for a history of alcohol and/or drug abuse as determined by the investigator

   H. Compliance:

   Subjects are excluded if they exhibit suspected or confirmed poor compliance in completing clinical study evaluations and/or clinical study required questionnaires.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2004-01-10 (Actual); Primary Completion 2005-03-11 (Actual); Study Completion 2005-03-11 (Actual)

PRIMARY OUTCOMES:
Evaluate subjects treated with ALX1-11 (no calcium supplementation) increase in BMD is less than those treated with ALX1-11 (receiving calcium supplementation). | 6 months
Primary efficacy variable is the percentage change from baseline of lumbar vertebral BMDmeasured by DXA. | 6 months

SECONDARY OUTCOMES:
BMC, | 6 months
vBMD, | 6 months
the incidence of clinical fractures, | 6 months
height, | 6 months
biochemical markers of bone turnover for subjects treated with ALX1-11 and receiving no calcium versus those receiving ALX1-11 with calcium supplementation. | 6 months
Adverse Events | 6 months
12 lead ECG changes | 6 months
Percentage change from baseline of lumbar vertebral BMC | 6 months
Percentage change from baseline of total hip BMD and BMC | 6 months
Percentage change from baseline in biochemical markers of bone turnover: 1) Bone formation: Serum BSAP and P1NP 2) Bone resorption: Serum CTx, urinary NTx | 6 months
Incidence of new and/or worsened vertebral (thoracic and lumbar) fractures | 6 months
Incidence of any clinical fractures (vertebral and/or non-vertebral) | 6 months
Incidence of hip fractures | 6 months
Incidence of clinical fractures other than hip, or thoracic or lumbar vertebrae | 6 months
Percentage change from baseline of trabecular volumetric BMD of spine as assessed by QCT (sub-study) | 6 months
Percentage change from baseline of trabecular volumetric BMD of hip as assessed by QCT (sub-study) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (27):
- United States (17):
  - 'Boling Clinical Trials, Rancho Cucamonga, California
  - 'Radiant Research - Lake Worth, Lake Worth, Florida
  - Odyssey Research/Bone Density of North Idaho, Coeur d'Alene, Idaho
  - 'The University of Chicago, Chicago, Illinois
  - 'University Hospital & Outpatient Center, Indianapolis, Indiana
  - 'Bethesda Health Research Center, Bethesda, Maryland
  - 'Michigan Bone & Mineral Clinic, Detroit, Michigan
  - Odyssey Research, North Platte, Nebraska
  - Creighton University School of Medicine, Omaha, Nebraska
  - 'New Mexico Clinical Research and Osteoporosis Center, Albuquerque, New Mexico
  - 'Odyssey Research Services, Bismarck, North Dakota
  - Michael J. Lillestol, Fargo, North Dakota
  - 'Odyssey Research Services, Minot, North Dakota
  - 'Radiant Research, Wyomissing, Pennsylvania
  - Odyssey Research/Avera United Clinic, Aberdeen, South Dakota
  - 'Brown Clinic, Watertown, South Dakota
  - 'Diabetes Center of the Southwest, Midland, Texas
- Argentina (2):
  - 'IDIM, Buenos Aires, BUE
  - 'Centro de Osteopatias Medicas, Capital Federal, CBA
- Mexico (8):
  - 'Hospital Clinical del Parque, Chihuahua City, CHIH
  - 'Hospital Angeles de las Lomas, Huixquilucan, EMEX
  - 'Hospital Aranda de la Parra, León, Guanajuato
  - 'OPD Hospital Civil de Guadalajara Dr. Juan I. Menchaca, Guadalajara, Jalisco
  - 'Hospital Civil de Belem, Guadalajara, Jalisco
  - 'Medica Monraz, Guadalajara, Jalisco
  - 'Instituto Mexicano de Investigacion Clinica, Mexico City, Mexico City
  - 'Hospital Universitario de Monterrey, Monterrey Nuevo Leon